CLINICAL TRIAL: NCT03506204
Title: The Pelvic Floor Muscle Function in Chinese Primipara, a One-year Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Liuzhou Maternity and Child Healthcare Hospital (Other); Maternity and Child Health Hospital of Dali (Unknown); Zhongshan People's Hospital, Guangdong, China (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Second Affiliated Hospital of Soochow University (Other); Maternity and Child Health Hospital of Changsha (Unknown); Henan Provincial People's Hospital (Other); Huaian Maternal and Child Health Care Hospital (Other); Hunan Provincial Maternal and Child Health Care Hospital (Other); The Fourth Hospital of Shijiazhuang (Other); Shenzhen Luohu District Maternity And Child Healthcare Hospital (Unknown); Second Affiliated Hospital of Wenzhou Medical University (Other); Hubei Shiyan People's Hospital (Unknown); Changzhi Maternity & Child Health Hospital (Other); Maternal and Child Health Care Hospital of Xinjiang Uygur Autonomous Region (Unknown); The First Hospital of Hebei Medical University (Other); Shen-Zhen City Maternity and Child Healthcare Hospital (Other); Dalian Medical University (Other); Maternity and Child Care Center of QinHuangDao City (Unknown); Chengdu Women's and Children's Central Hospital (Other); Shunyi Maternal and Children's Hospital of Beijing Children's Hospital (Unknown); Shandong Provincial Maternal and Child Health Care Hospital (Unknown); The People's Hospital of Leshan (Other); Hubei Maternal and Child Health Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: JS-1549
Record Dates: First submitted 2018-04-13; First posted 2018-04-24 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Pelvic Floor Muscle Weakness; Postpartum; Primiparity
Keywords: Pelvic floor muscle strength; Pelvic floor dysfunction; Postpartum; primipara

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is a prospective cohort study.The primiparas in six geographic regions of China are recruited to observe the natural recovery of pelvic floor muscle. The pelvic floor muscle function is evaluated at 6 weeks,3 months and 12 months after delivery.

DETAILED DESCRIPTION:
The primiparas in six geographic regions of China are recruited to observe the natural recovery of pelvic floor muscle.Evaluation of pelvic floor function is performed at 6 weeks, 3 months, 12 months after delivery. The modified Oxford Grading Scale and Levator ani testing are used to quantify PFM strength through vaginal palpation. Pelvic floor muscles strength, endurance, repetition,vaginal contraction pressure and the knack test are evaluated using a neuromuscular stimulation therapy system of PHENIX (Company: Vivaltis -Electronic Concept Lignon Innovation, Montpellier, France).

ELIGIBILITY:
Inclusion Criteria:

1. Women who give birth for the first time （Including vaginal delivery and cesarean section）
2. Term birth（37-42 weeks）
3. Single birth
4. Aged from 18 to 50
5. Plan to live locally for extended periods of time

Exclusion Criteria:

1. A history of incontinence before pregnancy
2. A history of fecal incontinence before pregnancy
3. Pelvic organ prolapse before pregnancy （prolapse out of the hymen ）
4. A history of abortion or induced labour over 16 weeks of pregnancy
5. Multiple pregnancy
6. The weight of the newborn is less than 2500g or more than 4000g
7. Precipitate labour
8. Operative vaginal delivery（obstetric forceps or vacuum extraction）
9. Laceration of perineum at least level III
10. Request for pelvic floor rehabilitation exercise（patients who have entered the group can not train the pelvic floor muscle）
11. Obesity （BMI before pregnancy over 25, BMI=weight (kg) / height square (m2) ）
12. Asthma
13. Long-term abdominal pressure（chronic cough for more than 1 months ，long-term constipation ect.）
14. Diabetes
15. Cotugno's disease
16. A history of pelvic floor surgery in the previous years

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Six geographic regions of China are needed to be covered, and more than 1-2 hospitals in each area should be included. The primipara are recruited while having their routine follow-up 6 weeks after delivery at the outpatient department in local hospitals.
Sampling Method: Probability Sample
Enrollment: 3120 (Estimated)
Dates: Start 2018-05-10 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum vaginal contraction pressure | Change from Baseline Maximum Vaginal Contraction Pressure in a year after delivery
  it is measured by manometry, range(80-150cmH2O). The higher values represent better outcomes.

SECONDARY OUTCOMES:
Pelvic floor muscle strength | change from baseline in a year after delivery
  The modified Oxford Grading Scale is used to quantify PFM strength through vaginal palpation.range(0-5).The higher values represent better outcomes.
Pelvic floor muscle strength（repetition） | change from baseline in a year after delivery
  Levator ani testing is used to quantify PFM strength.range(0-5).The higher values represent better outcomes.
Pelvic floor muscle contraction edurance | change from baseline in a year after delivery
  muscle contractions maintained for 0 s are defined as grade 0, 1 s as grade I, 2 s as grade II, 3 s as grade III, 4 s as grade IV, and 5 s or longer as grade V. Normal muscles can maintain the contraction for 5 s.range(0-5s).The higher values represent better outcomes.
the knack test | change from baseline in a year after delivery
  a voluntary PFM contraction before or during coughing.That the contraction could be performed represents normal.
vaginal rest pressure | change from baseline in a year after delivery
  measure when no vaginal contraction by manometry. range(25-50 cmH2O). the lower and the higher values represent abnormal outcomes.
Condition of stress urinary incontinence | change from baseline in a year after delivery
  Ingelman-Sundberg classification is used according to the clinical symptoms of urinary incontinence, divided into mild, moderate and severe.
pelvic organ prolapse quantification(POP-Q) | change from baseline in a year after delivery
  POP-Q is measured when maximum valsalva.range(0-4). stage 0 represents normal.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, MD, Principal Investigator — Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences, Beijing, Beiing, China